CLINICAL TRIAL: NCT06906484
Title: Diagnostic Value of Systematic Echocardiography in the Cardiovascular Screening of Amateur Football Referees
Brief Title: Systematic Transthoracic Echocardiographic Screening in Amateur Football Referees
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: REF-TTE
Record Dates: First submitted 2025-03-21; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Sreening; Soccer Referees
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: echocardiography — analyse echocardiographic reports on cardiac abnomalies

SUMMARY:
This retrospective study aims to evaluate the prevalence of cardiac abnormalities detected by transthoracic echocardiography (TTE) in amateur football referees as part of a systematic cardiovascular screening program.

DETAILED DESCRIPTION:
cardiovasculaire screening of athletes and sports officials is essential for preventing sudden cardiac death during physical activity. In 2019, the French Football Federation (FFF) introduced mandatory transthoracic echocardiography (TTE) for amateur referees over 18 years old, to improve early detection of cardiovascular abnormalities.

This retrospective observational study investigates the diagnostic value of systematic TTE in detecting structural or functional cardiac anomalies among adult amateur referees affiliated with the Normandy Football League.

The primary objective is to estimate the prevalence of cardiac abnormalities diagnosed by TTE in this population. The secondary objectives include identifying the prevalence of cardiovascular risk factors (CVRFs), and describing the abnormalities found during the medical evaluation

ELIGIBILITY:
Inclusion Criteria:

Male amateur football referees, aged ≥18 Affiliated with the Normandy Football League Completed a baseline TTE No known pre-existing cardiac disease Complete medical records available

Exclusion Criteria:

Referees under 18 or in training status History of cardiovascular disease Incomplete medical file

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes amateur football referees affiliated with the Normandy Football League (France) who actively officiated since the 2022 season.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of structural or functional abnormalities detected by TTE | At the baseline
  The primary outcome is the proportion of participants presenting with significant structural or functional cardiac abnormalities detected by resting transthoracic echocardiography performed as part of the mandatory cardiovascular screening for amateur football referees.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de CAEN, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided